CLINICAL TRIAL: NCT05313984
Title: Optimization of Therapy Resistant LUTS (OptiLUTS) Part C: the Development of a Symptom Assessment Tool in Sacral Neuromodulation: a Prospective Single Centre Study.
Brief Title: OptiLUTS Part C: the Development of a Symptom Assessment Tool in Sacral Neuromodulation.
Acronym: OptiLUTS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: EC2018/0244
Record Dates: First submitted 2022-03-03; First posted 2022-04-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Overactive Bladder Syndrome; Urinary Retention; Dysfunctional Voiding; Fecal Incontinence; Fowler Syndrome
Keywords: Sacral neuromodulation
MeSH Terms: conditions — Urinary Retention; Fecal Incontinence; Fowler Christmas Chapple syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients planned for the 2-staged tined-lead procedure.: Patients with the following indications:
  * Overactive bladder without urgency urinary incontinence.
  * Overactive bladder with urgency urinary incontinence.
  * Non-obstructive urinary retention.
  * Dysfunctional voiding or Fowler Syndrome.
  * Fecal incontinence.
  Interventions: Device: Sacral neuromodulation

INTERVENTIONS:
Device: Sacral neuromodulation — Sacral neuromodulation: the 2-staged tined lead procedure. (Interstim II therapy, Medtronic).
  Stage I: Placement of a tined-lead electrode. 2 - 4 weeks test phase. Stage II: Placement of an implantable pulse generator.
  Other Names: SNM

SUMMARY:
Sacral neuromodulation (SNM) is a two-staged 2nd-line therapy for therapy-resistant LUTS and fecal incontinence. Currently, the assessment of symptoms at baseline and after stage I is directed towards a discipline related evaluation. The OptiLUTS trial strives for a more holistic approach, taking all pelvic floor dysfunctions into account.

A holistic assessment tool will be developed and SNM-care pathway will be set-up.

DETAILED DESCRIPTION:
A prospective single centre trial is set up. Patients planned for the two-staged tined lead procedure are enrolled.

Bladder and bowel diaries and patient reported outcome measures (PROMS) will be collected at baseline and in between stage I and stage II, and PROMS at one month, 6 months and 12 months after definitive implant.

Phase I Step 1: The current implant rate, true success rate, outcomes and false positive rate will be measured.

Step 2: Development of a holistic symptom assessment tool. Phase II Implementation of the SNM care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years presenting with one or more of the following indications: Urinary urgency frequency with or without urinary incontinence (OAB dry or wet), non-obstructive urinary retention, dysfunctional voiding with post void residual volume, faecal incontinence and mixed incontinence
* Refractory to conservative treatment (i.e. Lifestyle changes, behavioural modification, pelvic floor muscle training, biofeedback) and refractory to pharmacological treatment.

Exclusion Criteria:

* Neurogenic bladder.
* Anal sphincter damage more than 120
* Abnormal sacral anatomy
* Mentally or physically disabled patients not capable to handle a patient programmer device.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for pelvic organ dysfunctions to the Urology department (UD) and Colorectal Surgery department (CRD) of the Ghent University Hospital and scheduled for a staged SNM procedure using InterstimTM II therapy (Medtronic, Minneapolis, MN) were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Implantation ratio | Through study completion, an average of 3 years
  Proportion of number of patients who received a definitive implant.
True success ratio | Through study completion, an average of 3 years
  Proportion of patients showing both objective (ObS) and subjective success (SS) during the test phase of SNM.
False positive ratio | One month after definitive implant.
  Proportion of patients with discontinued SS although having true success during test phase.

SECONDARY OUTCOMES:
Explantation ratio | Within 12 months after definitive implant.
  Proportion of patients explanted.
Revision ratio | Within 12 months after definitive implant.
  Proportion of patients that received a revision.
Absolute change in diary variables. | Up to 4 weeks, depending on the duration of the test phase.
  Test phase compared to baseline. (Different for each indication).
Evolution of PROM scores over time. | At 12 months follow-up.
  Total PROM scores, based on questionnaires, baseline compared to scores at during the test phase vs. at 1 month, at 6 months and at 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Everaert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Department of Urology, Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghijselings L, Verbakel I, Bou Kheir G, Van de Putte D, Herve F, Goessaert AS, Pauwaert K, Beeckman D, Ooms M, Everaert K. Symptom Assessment of Candidates for Sacral Neuromodulation Therapy With Urologic and Colorectal Conditions: Time for a Holistic Approach? Results and Findings From a Prospective Single-Center Study. Neuromodulation. 2025 Jul;28(5):847-857. doi: 10.1016/j.neurom.2024.04.009. Epub 2024 Jun 6. PMID 38842955